CLINICAL TRIAL: NCT01336569
Title: Safety and Efficacy of Using the Travoprost/Timolol Fixed Combination (DuoTrav®) in Patients With Open-Angle Glaucoma or Uncontrolled Ocular Hypertension by Beta-blocker Monotherapy (Timolol 0.5%)
Brief Title: Safety and Efficacy of Changing to DuoTrav in Patients Uncontrolled on Timolol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMA-09-26
Record Dates: First submitted 2011-04-14; First posted 2011-04-18 (Estimated); Results first posted 2013-07-08 (Estimated); Last update posted 2013-07-08 (Estimated); Status verified 2013-05

CONDITIONS: Glaucoma
Keywords: Primary Open-Angle Glaucoma; Ocular Hypertension; Pigment Dispersion Glaucoma; IOP
MeSH Terms: conditions — Glaucoma; Glaucoma, Open-Angle; Ocular Hypertension | interventions — Travoprost; Timolol; Duotrav

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DuoTrav (Experimental): Travoprost 0.004%/timolol maleate 0.5% fixed combination, one drop to the study eye nightly for up to 6 weeks
  Interventions: Drug: Travoprost 0.004%/timolol maleate 0.5% fixed combination

INTERVENTIONS:
Drug: Travoprost 0.004%/timolol maleate 0.5% fixed combination
  Other Names: DuoTrav

SUMMARY:
The purpose of this study was to assess the safety and intraocular pressure (IOP)-lowering efficacy of changing to DuoTrav® from prior timolol 0.5% monotherapy in participants with open-angle glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ocular hypertension, primary open-angle glaucoma or pigmentary glaucoma;
* Intraocular pressure (IOP) of between 19 to 35 mmHg at any time of the day in at least one eye (designated as the study eye);
* On a stable medication regimen for IOP reduction one week prior to the screening visit;
* Best corrected visual acuity better than 20/200 (Snellen) or 1.0 (logMAR) in each eye;
* Sign informed consent;
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Known medical history of allergy, hypersensitivity or low tolerance to any of the components of DuoTrav®;
* Any abnormality that would preclude the reliable performance of applanation tonometry in either eye;
* Infection in either eye;
* Conventional or laser intraocular surgery in either eye 3 months prior to screening visit;
* Risk for visual field or visual acuity worsening, in the opinion of the investigator;
* Women of childbearing potential;
* Pregnant or lactating women;
* Any condition that, in the opinion of the principal investigator, could interfere with participation in the study, or that could present a risk to the participant.
* Participation in another clinical study within 30 days before the screening visit;
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-02; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abayomi Ogundele, PharmD, Study Director — Alcon Research
Locations (1):
- Contact Alcon Call Center for Trial Locations, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited and enrolled from 4 study centers located in Brazil.
Pre-assignment Details: Of the 50 enrolled, 1 participant did not meet inclusion/exclusion criteria and was exited from the study prior to receiving study product. This reporting group includes all participants who received study product.
Period: Overall Study
Arm/Group | DuoTrav
Started | 49
Completed | 45
Not Completed | 4
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Population: This reporting group includes all participants who received study product.
Arm/Group | DuoTrav
Number analyzed (Participants) | 49
Age Continuous [Mean (Standard Deviation); unit: years] | 63.3 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 13
Region of Enrollment [Number; unit: participants]
  Brazil | 49

OUTCOME MEASURES:

1. Primary Outcome: Mean Intraocular Pressure (IOP) Change at the Final Visit From Baseline (Prior Beta-blocker Monotherapy)
Description: As measured by Goldmann applanation tonometry. High IOP (outside the normal range) can be a risk factor for developing glaucoma or glaucoma progression (leading to optic nerve damage). A more negative change indicates a greater amount of improvement.
Time Frame: Baseline, up to 6 weeks
Population: Intent-to-Treat (ITT): All participants who received study medication and had at least one on-therapy study visit.
Measure: Mean (Standard Deviation); unit: millimeters mercury (mmHg)
Arm/Group | DuoTrav
Number analyzed (Participants) | 45
millimeters mercury (mmHg) | -5.0 (3.6)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study.
Description: This reporting group includes all participants who received study product.
Arm/Group | DuoTrav
Serious Adverse Events (participants affected / at risk) | 1/49
Other Adverse Events (participants affected / at risk) | 0/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DuoTrav (N=49)
Enterorrhagia (Gastrointestinal disorders) | 1 — Not related

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.